CLINICAL TRIAL: NCT03868709
Title: Impact of Prophylactic Penehyclidine Hydrochloride Inhalation on Long-term Outcome in High-risk Patients: 3-year Follow-up of a Randomized Controlled Trial
Brief Title: Prophylactic Penehyclidine Hydrochloride Inhalation and 3-year Outcome After Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018[213]
Record Dates: First submitted 2019-03-03; First posted 2019-03-11 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Complications; Long-term Outcome
Keywords: Postoperative pulmonary complications; Penehyclidine Hydrochloride; High risk patients; Postoperative period; Long-term outcome
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Penehyclidine group (Experimental): Penehyclidine inhalation is administered (penehyclidine hydrochloride 0.5 mg/0.5 ml + normal saline 5.5 ml) once every 12 hours from the night before surgery till the second day after surgery. The total number of inhalation is seven times. Study drug inhalation is performed with the high-flow oxygendriven method for the non-intubated patients or with the atomizing inhalation device of ventilator for the intubated patients.
  Interventions: Drug: Penehyclidine inhalation
- Placebo group (Placebo Comparator): Placebo inhalation is administered by inhalation (water for injection 0.5 ml + normal saline 5.5 ml ) once every 12 hours from the night before surgery till the second day after surgery. The total number of inhalation is seven times. Study drug inhalation will be performed with the high-flow oxygen-driven method for the non-intubated patients or with the atomizing inhalation device of ventilator for the intubated patients.
  Interventions: Drug: Placebo inhalation

INTERVENTIONS:
Drug: Penehyclidine inhalation — Penehyclidine inhalation is administered by inhalation (penehyclidine hydrochloride 0.5 mg/0.5 ml, mixed with normal saline 5.5 ml) once every 12 hours from the night before surgery till the second day after surgery. The total number of inhalation is seven times. Study drug inhalation is performed with the high-flow oxygen-driven method for the non-intubated patients or with the atomizing inhalation device of ventilator for the intubated patients
  Arms: Penehyclidine group
Drug: Placebo inhalation — Placebo inhalation is administered by inhalation (water for injection 0.5 ml, mixed with normal saline 5.5 ml) once every 12 hours from the night before surgery till the second day after surgery. The total number of inhalation is seven times. Study drug inhalation is performed with the high-flow oxygendriven method for the non-intubated patients or with the atomizing inhalation device of ventilator for the intubated patients.
  Arms: Placebo group

SUMMARY:
Postoperative pulmonary complications (PPCs) are major causes of postoperative morbidity, mortality, and prolonged hospital stay.The incidence of PPCs may be as high as 41% to 75% in high-risk patients. Bronchodilator is frequently used in high-risk patients to prevent PPCs. Penehyclidine is a new anticholinergic agent which selectively block M1 and M3 receptors. A previous randomized controlled trial tested the effect of prophylactic penehyclidine inhalation on the incidence of PPCs in high-risk patients. The purpose of this 3-year follow-up study is to investigate whether prophylactically penehyclidine hydrochloride inhalation can affect the 3-year outcomes of patients recruited in the previous randomized controlled trial.

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPCs) are major causes of postoperative morbidity, mortality, and prolonged hospital stay. The incidence of PPCs was found to vary from 2 to 19%, but this rate may be as high as 41 to 75% in patients after intrathoracic and intraabdominal surgery. According to Canet's model, the predicted incidence of PPCs in high-risk patients (ARISCAT risk index ≥45 points) is 42.1%.

Use of effective strategies to prevent PPCs is essential for those high-risk patients. As a bronchodilator, anticholinergic inhalation may be helpful. Studies showed that, in high-risk patients undergoing intrathoracic surgery, airway resistance is increased due to bronchial hyperresponsiveness, which increased the risk of PPCs. Inhalation of anticholinergic bronchodilator can reduce the activity of vagus nerve and relieve high airway resistance, which may decrease the risk of bronchospasm and other PPCs. It has been shown that M1, M3-receptor selective blockers have better effects than β2-receptor activator in dilating bronchia.

Penehyclidine hydrochloride is a new anticholinergic agent, which selectively blocks M1 and M3 receptors. Preclinical studies found that it also has anti-inflammation effects. In a pilot study of the investigators, prophylactic inhalation of penehyclidine decreased the incidence of bronchospasm and the use of aminophylline in elderly patients after long-duration surgery. In a previous randomized controlled trial, 864 high-risk patients were recruited and randomized to receive prophylactic inhalation of either penehyclidine or placebo.

The investigators hypothesize that prophylactically penehyclidine hydrochloride inhalation may improve long-term outcomes in this patient population by reducing PPCs. The purpose of this 3-year follow-up study is to investigate whether prophylactically penehyclidine hydrochloride inhalation can affect the 3-year outcomes in high-risk patients recruited in the previous randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 50 years or over;
2. Scheduled to undergo open or laparoscope assisted upper abdominal or intrathoracic surgery;
3. The expected duration of surgery is 2 hours or longer;
4. Identified at high risk of PPCs according to the ARISCAT risk score (ARISCAT predictive score ≥45).

Exclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical classification ≥ IV or the expected survival duration ≤ 24 h;
2. Preoperative history of prostatic hypertrophy or glaucoma;
3. History of myocardial infarction, severe heart dysfunction (New York Heart Association functional classification ≥ 3) or tachyarrhythmia within one year;
4. Inhalation of β2-receptor activator, M-receptor blockers and/or glucocorticoids within one month before surgery;
5. Severe renal dysfunction (requirement of renal replacement therapy) or severe hepatic dysfunction (Child-Pugh grade C);
6. History of acute stroke within three months before surgery;
7. Refuse to participate in the study or unable to cooperate with the inhalation therapy;
8. Participation in other clinical trial during the last month or within the six half-life periods of the study drug used in the last trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Duration of overall survival within 3 years after surgery | From the day of surgery until the end of the 3rd year after surgery
  Duration of overall survival within 3 years after surgery

SECONDARY OUTCOMES:
Survival rates at different timepoints after surgery | At the end of the 1st, 2nd, and 3rd year after surgery
  Survival rates at different timepoints after surgery
Duration of recurrence-free survival within 3 years after surgery | From the day of surgery until the end of the 3rd year after surgery
  Duration of recurrence-free survival within 3 years after surgery for primary cancer
Ocurrence of new-onset diseases during the 3-year period after surgery | From the day of surgery until the end of the 3rd year after surgery
  New-onset diseases indicate those that occurred during the 3-year period after surgery and required medical therapy, such as acute myocardial infarction, stroke, new cancer, etc.
Cognitive function of 3-year survivors | Assessed at the end of the 3rd year after surgery
  Cognitive function is assessed with the Telephone Interview for Cognitive Status-Modified (TICS-m)
The quality of life in 3-year survivors | Assessed at the end of the 3rd year after surgery
  The quality of life is assessed with the World Health Organization Quality of Life-BREF (WHOQOL-BREF)
The quality of life in 3-year survivors with chronic pulmonary disease | Assessed at the end of the 3rd year after surgery
  The quality of life is assessed with the St. George's Respiratory Questionnaire (SGRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher BW, Majumdar SR, McAlister FA. Predicting pulmonary complications after nonthoracic surgery: a systematic review of blinded studies. Am J Med. 2002 Feb 15;112(3):219-25. doi: 10.1016/s0002-9343(01)01082-8. PMID 11893349
- [Background] Khuri SF, Henderson WG, DePalma RG, Mosca C, Healey NA, Kumbhani DJ; Participants in the VA National Surgical Quality Improvement Program. Determinants of long-term survival after major surgery and the adverse effect of postoperative complications. Ann Surg. 2005 Sep;242(3):326-41; discussion 341-3. doi: 10.1097/01.sla.0000179621.33268.83. PMID 16135919
- [Background] Sabate S, Mazo V, Canet J. Predicting postoperative pulmonary complications: implications for outcomes and costs. Curr Opin Anaesthesiol. 2014 Apr;27(2):201-9. doi: 10.1097/ACO.0000000000000045. PMID 24419159
- [Background] Wu CL, Hurley RW, Anderson GF, Herbert R, Rowlingson AJ, Fleisher LA. Effect of postoperative epidural analgesia on morbidity and mortality following surgery in medicare patients. Reg Anesth Pain Med. 2004 Nov-Dec;29(6):525-33; discussion 515-9. doi: 10.1016/j.rapm.2004.07.002. PMID 15635510
- [Background] Matot I, Oppenheim-Eden A, Ratrot R, Baranova J, Davidson E, Eylon S, Peyser A, Liebergall M. Preoperative cardiac events in elderly patients with hip fracture randomized to epidural or conventional analgesia. Anesthesiology. 2003 Jan;98(1):156-63. doi: 10.1097/00000542-200301000-00025. PMID 12502992
- [Background] Melduni RM, Koshino Y, Shen WK. Management of arrhythmias in the perioperative setting. Clin Geriatr Med. 2012 Nov;28(4):729-43. doi: 10.1016/j.cger.2012.08.006. PMID 23101581
- [Background] Antoniou SA, Antoniou GA, Koch OO, Kohler G, Pointner R, Granderath FA. Laparoscopic versus open obesity surgery: a meta-analysis of pulmonary complications. Dig Surg. 2015;32(2):98-107. doi: 10.1159/000371749. Epub 2015 Mar 3. PMID 25765889
- [Background] Lawrence VA, Hilsenbeck SG, Mulrow CD, Dhanda R, Sapp J, Page CP. Incidence and hospital stay for cardiac and pulmonary complications after abdominal surgery. J Gen Intern Med. 1995 Dec;10(12):671-8. doi: 10.1007/BF02602761. PMID 8770719
- [Background] Khan NA, Quan H, Bugar JM, Lemaire JB, Brant R, Ghali WA. Association of postoperative complications with hospital costs and length of stay in a tertiary care center. J Gen Intern Med. 2006 Feb;21(2):177-80. doi: 10.1111/j.1525-1497.2006.00319.x. PMID 16606377
- [Background] Kor DJ, Warner DO, Alsara A, Fernandez-Perez ER, Malinchoc M, Kashyap R, Li G, Gajic O. Derivation and diagnostic accuracy of the surgical lung injury prediction model. Anesthesiology. 2011 Jul;115(1):117-28. doi: 10.1097/ALN.0b013e31821b5839. PMID 21694510
- [Background] Ramachandran SK, Nafiu OO, Ghaferi A, Tremper KK, Shanks A, Kheterpal S. Independent predictors and outcomes of unanticipated early postoperative tracheal intubation after nonemergent, noncardiac surgery. Anesthesiology. 2011 Jul;115(1):44-53. doi: 10.1097/ALN.0b013e31821cf6de. PMID 21552116
- [Background] Smith PR, Baig MA, Brito V, Bader F, Bergman MI, Alfonso A. Postoperative pulmonary complications after laparotomy. Respiration. 2010;80(4):269-74. doi: 10.1159/000253881. Epub 2009 Oct 28. PMID 19864881
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Thomsen T, Villebro N, Moller AM. Interventions for preoperative smoking cessation. Cochrane Database Syst Rev. 2014 Mar 27;2014(3):CD002294. doi: 10.1002/14651858.CD002294.pub4. PMID 24671929
- [Background] Kroenke K, Lawrence VA, Theroux JF, Tuley MR. Operative risk in patients with severe obstructive pulmonary disease. Arch Intern Med. 1992 May;152(5):967-71. PMID 1580723
- [Background] Celli BR. Perioperative respiratory care of the patient undergoing upper abdominal surgery. Clin Chest Med. 1993 Jun;14(2):253-61. PMID 8519171
- [Background] Hulzebos EH, Smit Y, Helders PP, van Meeteren NL. Preoperative physical therapy for elective cardiac surgery patients. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD010118. doi: 10.1002/14651858.CD010118.pub2. PMID 23152283
- [Background] Yan T, Wang D. [Effects of penehyclidine inhalation on postoperative pulmonary complications of elderly patients after long-duration surgery]. Zhonghua Yi Xue Za Zhi. 2014 Jan 14;94(2):122-6. Chinese. PMID 24721352
- [Background] Wu GM, Mou M, Mo LQ, Liu L, Ren CH, Chen Y, Zhou J. Penehyclidine hydrochloride postconditioning on lipopolysaccharide-induced acute lung injury by inhibition of inflammatory factors in a rodent model. J Surg Res. 2015 May 1;195(1):219-27. doi: 10.1016/j.jss.2014.12.018. Epub 2014 Dec 17. PMID 25577143